CLINICAL TRIAL: NCT06109402
Title: Perioperative Immunotherpay Versus Adjuvant Immunotherapy for Resectable Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-019
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Stage II-IIIB(N2) Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; 130-nm albumin-bound paclitaxel; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative immunotherapy (Experimental): In this arm, patients will receive neoadjuvant immunochemotherapy and adjuvant immunotherapy.
  Interventions: Drug: TQB2450; Drug: Carboplatin; Drug: Pemetrexed; Drug: Nab-paclitaxel; Procedure: Surgery
- Adjuvant immunotherapy (Experimental): In this arm, patients will receive adjuvant immunochemothrapy and immunotherapy
  Interventions: Drug: TQB2450; Drug: Carboplatin; Drug: Pemetrexed; Drug: Nab-paclitaxel; Procedure: Surgery

INTERVENTIONS:
Drug: TQB2450 — Specified dose on specified days
Drug: Carboplatin — Specified dose on specified days
Drug: Pemetrexed — Specified dose on specified days
Drug: Nab-paclitaxel — Specified dose on specified days
Procedure: Surgery — Surgery for II-IIIB (N2) non-small cell lung cancer

SUMMARY:
For resectable non-small cell lung cancer, neoadjuvant immunochemotherapy plus adjuvant immunotherapy or adjuvant immunochemotherapy is usually used in clinical practice. However, it is unclear whether therapeutic strategy is superior. This trial aims to compare the efficacy and safety of these two strategies.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form.
2. Aged 18 ≥ years.
3. Histological or cytological diagnosis of NSCLC by needle biopsy, and stage II-IIIB (N2) confirmed by imageological examinations (CT, PET-CT or EBUS).
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
5. Life expectancy is at least 12 weeks.
6. At least 1 measurable lesion according to RECIST 1.1.
7. Patients with good function of other main organs (liver, kidney, blood system, etc.)
8. Patients with lung function can tolerate surgery;
9. Without systematic metastasis (including M1a, M1b and M1c);
10. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of immunotherapy (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
11. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of immunotherapy (whichever is later).

Exclusion Criteria:

1. Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
2. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
3. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
4. Participants who are allergic to the test drug or any auxiliary materials;
5. Participants with Interstitial lung disease currently;
6. Participants with active hepatitis B, hepatitis C or HIV;
7. Pregnant or lactating women;
8. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
9. Participated in another therapeutic clinical study;
10. Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
3-year event-free survival (EFS) rate | Up to 48 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:
  the appearance of one or more new lesions is also considered progression).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 6 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the neoadjuvant therapy. Only patients with measurable lesions at baseline will be analyzed.
Pathological complete response (pCR) | Up to 8 months
  pCR is defined as the proportion of participants who have achieved complete pathologic response (on routine hematoxylin and eosin staining, tumors with no viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.
Major pathologic response (MPR) | Up to 8 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.
Event-free survival (EFS) | Up to 72 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:
  the appearance of one or more new lesions is also considered progression).
Overall survival (OS) | Up to 72 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
5-year event-free survival (EFS) rate | Up to 72 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:
  the appearance of one or more new lesions is also considered progression).
5-year overall survival (OS) | Up to 72 months
  OS is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Adverse event rate | Up to 36 months
  It is defined as the frequency of severe adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.
Health related quality of life (HRQol) | Up to 36 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.